CLINICAL TRIAL: NCT02962895
Title: Study of Safety and Efficacy of Multiple VAY736 Doses in Patients With Moderate to Severe Primary Sjogren's Syndrome (pSS)
Brief Title: Safety and Efficacy of VAY736 in Patients With Primary Sjogren's Syndrome (pSS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAY736A2201
Record Dates: First submitted 2016-11-03; First posted 2016-11-15 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Primary Sjogren Syndrome
Keywords: Sjogren; VAY736; ianalumab; pSS
MeSH Terms: interventions — ianalumab

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, placebo-controlled, multicenter, parallel-group trial which planned to enroll approximately 180 patients with moderate to severe primary Sjögren's syndrome. The study was divided into 4 study periods:
  Period 1: 4-week Screening to assess patient eligibility.
  Period 2: 24-week Blinded treatment period.
  Period 3: An extended blinded treatment period of 28 weeks. After Week 24 assessments, patients in the ianalumab 300 mg arm were re-randomized in a 1:1 ratio to either continue on ianalumab 300 mg s.c. q4w or switch to matching placebo up to Week 52.
  Period 4: Post-treatment safety follow-up period. Patients who prematurely discontinued the study treatment at any time point or completed the treatment as planned entered the safety follow-up period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VAY736 dose 1 - 5mg (Experimental): VAY736 low
  Interventions: Biological: VAY736
- VAY736 dose 2 - 50mg (Experimental): VAY736 medium
  Interventions: Biological: VAY736
- VAY736 dose 3 - 300 mg (Experimental): VAY736 high
  Interventions: Biological: VAY736
- Placebo (Placebo Comparator): Placebo control
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAY736 — VAY736
  Other Names: Ianalumab
  Arms: VAY736 dose 1 - 5mg; VAY736 dose 2 - 50mg; VAY736 dose 3 - 300 mg
Other: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the dose-response relationship of VAY736 for key efficacy and safety parameters

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multicenter, parallel-group trial that was divided into 4 study periods.

Period 1: A screening period of 4 weeks to assess patient eligibility. Patients could be re-screened only once, and no study-related re-screening procedure could be performed prior to written re-consent by the patient.

Period 2: A blinded treatment period of 24 weeks. At baseline, eligible patients were randomized to one of three ianalumab dose arms (VAY736 5 mg, 50 mg or 300 mg s.c.) or a placebo arm (placebo s.c.). Blinded study drug was administered every four weeks (q4w) for a 24-week period.

Except for Japan, randomization was stratified by baseline ESSDAI score (<10 or ≥10 based on weighted scores). Separate blocks of randomization numbers were generated for patients in Japan versus the other countries participating to ensure that Japanese patients were equally distributed across all treatment groups in the study.

The primary endpoint was assessed at the end of Period 2 (Week 24). Treatment assignment in Period 2 remained double-blinded until the end of Period 3.

Period 3: An extended blinded treatment period of 28 weeks. After Week 24 assessments, patients in the ianalumab 300 mg arm were re-randomized in a 1:1 ratio to either continue on ianalumab 300 mg s.c. q4w or switch to matching placebo up to Week 52. Patients who received placebo during Period 2 were switched to ianalumab 150 mg s.c q4w up to Week 52. Patients who received 5 mg and 50 mg s.c. in Period 2 proceeded directly to safety follow-up (Period 4). Treatment assignment in Period 3 remained double-blinded.

Period 4: A post-treatment safety follow-up period. Patients who prematurely discontinued the study treatment at any time point or completed the treatment as planned entered the safety follow-up period. The minimum required duration of follow-up in the study was 20 weeks from the last administration of the study treatment (mandatory follow-up). The maximum duration of the follow-up was 2 years from the last dose of the study treatment, and it was defined by the level of recovery of CD19+ B-cells: conditional follow up (with reduced visit frequency) until CD19+ B-cell levels return to at least 80% of baseline or 50 cells/µL, whichever occurred first. Patients who had not yet recovered their B-cell counts two years after last ianalumab dosing were discharged from the study and had undergone their End of Study (EoS) visit. Patients who were treated with another immunomodulatory or immunosuppressive treatment (e.g., azathioprine, cyclophosphamide, high dose glucocorticosteroids) after completion of the minimum 20-week safety follow-up period were excluded from further safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled revised American European Consensus Group criteria for pSS
* Seropositive at screening for anti-Ro/SSA antibodies
* Screening ESSDAI value >=6 scored from 7 domains: articular, cutaneous, glandular, lymphoadenopathy, constitutional, biologic and hematologic.

Exclusion Criteria:

* Secondary Sjogren's syndrome
* Use of other investigational drugs
* Active viral, bacterial or other infections
* Positive hepatitis B, hepatitis C, HIV or tuberculosis test results at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (52):
- United States (9):
  - Integral Rheumatology and Immunology Specialists IRIS, Plantation, Florida
  - Indiana Univ School of Dentistry, Indianapolis, Indiana
  - The John Hopkins Jerome L Greene Sjogren, Baltimore, Maryland
  - Tufts School of Dental Medicine, Boston, Massachusetts
  - AAIR Research Center, Rochester, New York
  - UPMC, Pittsburgh, Pennsylvania
  - Advanced Rheumatology and Arthritis Wellness Center, Wexford, Pennsylvania
  - Baylor College Of Medicine, Houston, Texas
  - First Outpatient Research Unit, San Antonio, Texas
- Argentina (3):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Graz, Austria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Santiago, Chile
- France (2):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Lille
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (3):
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Udine, UD
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Rotterdam, South Holland, Netherlands
- Novartis Investigative Site, Lublin, Poland
- Portugal (3):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (2):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Spain (3):
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Barcelona
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Southend

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bowman SJ, Fox R, Dorner T, Mariette X, Papas A, Grader-Beck T, Fisher BA, Barcelos F, De Vita S, Schulze-Koops H, Moots RJ, Junge G, Woznicki JN, Sopala MA, Luo WL, Hueber W. Safety and efficacy of subcutaneous ianalumab (VAY736) in patients with primary Sjogren's syndrome: a randomised, double-blind, placebo-controlled, phase 2b dose-finding trial. Lancet. 2022 Jan 8;399(10320):161-171. doi: 10.1016/S0140-6736(21)02251-0. Epub 2021 Nov 30. PMID 34861168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 190 Patients were enrolled from 56 centers in 19 countries.
Pre-assignment Details: Patients who were in the placebo arm in Period 2 were switched to VAY736 - 150mg s.c. administration every 4 weeks in Period 3.
  At the end of Period 2, patients from the VAY736 300mg every 4 weeks arm were re-randomized to either i) double-blind VAY736 300mg every 4 weeks or ii) double-blind placebo every four weeks. All other patients proceeded directly from Period 2 to Period 4 (Safety Follow-Up).
Groups:
- Placebo (Up to Week 24); VAY736 - 5 mg (Up to Week 24); VAY736 - 50 mg (Up to Week 24); VAY736 - 300 mg (Up to Week 24): Period 2 (Double blind Placebo s.c. administration every 4 weeks (q4w) for a 24-week period)
- VAY736 - 150 mg: Placebo patients in Period 2 switched to VAY736 - 150 mg s.c. administration every 4 weeks in Period 3 (Period 3 = 28 weeks)
- VAY736 300 mg - Placebo: VAY736 300 mg patients in Period 2 re-randomized to Placebo every 4 weeks in Period 3 (Period 3 = 28 weeks)
- VAY736 300 mg - VAY736 300 mg: VAY736 300 mg patients in Period 2 re-randomized to VAY736 300 mg every 4 weeks in Period 3 (Period 3 = 28 weeks)
Period: Period 2 (Randomized Set: Up to Week 24)
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | VAY736 - 150 mg | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Set (SAF)) | 49 | 47 | 47 | 47 | 0 | 0 | 0
Completed | 47 | 42 | 43 | 46 | 0 | 0 | 0
Not Completed | 2 | 5 | 4 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — New therapy for indication | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3 (Randomized Set / Weeks: 24-52)
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | VAY736 - 150 mg | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Started | 0 | 0 | 0 | 0 | 47 | 22 | 21
Completed | 0 | 0 | 0 | 0 | 42 | 22 | 17
Not Completed | 0 | 0 | 0 | 0 | 5 | 0 | 4
Not completed — Patient/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 4 (Safety Follow-Up)
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | VAY736 - 150 mg | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Started | 2 | 47 | 47 | 4 | 46 | 22 | 20
Completed | 2 | 41 | 43 | 1 | 42 | 20 | 20
Not Completed | 0 | 6 | 4 | 3 | 4 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — New therapy for indication | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of informed consent | 0 | 3 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 1 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | Total
Number analyzed (Participants) | 49 | 47 | 47 | 47 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (12.44) | 52.5 (13.64) | 51.0 (11.12) | 49.1 (15.41) | 50.9 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 41 | 46 | 180
  Male | 2 | 1 | 6 | 1 | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 4 | 3 | 10 | 5 | 22
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 44 | 42 | 37 | 42 | 165
  Unknown | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in ESSDAI Score at Week 24
Description: The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) instrument contains 12 organ-specific domains contributing to disease activity. For each domain, features of disease activity are scored in 3 or 4 levels according to their severity. These scores are then summed across the 12 domains in a weighted manner to provide the total score ranging 0-123. Higher scores on the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states. A negative change from baseline indicates improvement in disease status.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale | -6.39 (0.808) | -5.64 (0.850) | -6.93 (0.836) | -8.30 (0.828)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo; Test type: Superiority; p = 0.5161, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.75, 95% CI 2-sided [-1.52 to 3.02]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo; Test type: Superiority; p = 0.6332, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -0.55, 95% CI 2-sided [-2.80 to 1.71]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo; Test type: Superiority; p = 0.0921, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -1.92, 95% CI 2-sided [-4.15 to 0.32]

2. Secondary Outcome: Least Squares Mean Change From Baseline in ESSDAI Score at Weeks 4, 8, 12, and 16
Description: as for outcome 1
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Week 4: number analyzed (Participants) | 49 | 46 | 46 | 45
  Week 4 | -3.73 (0.626) | -2.28 (0.661) | -3.37 (0.638) | -4.53 (0.651)
  Week 8: number analyzed (Participants) | 47 | 46 | 44 | 46
  Week 8 | -4.13 (0.704) | -4.65 (0.733) | -4.73 (0.720) | -6.38 (0.717)
  Week 12: number analyzed (Participants) | 49 | 44 | 45 | 46
  Week 12 | -5.45 (0.721) | -4.89 (0.762) | -5.69 (0.739) | -6.64 (0.739)
  Week 16: number analyzed (Participants) | 48 | 46 | 46 | 46
  Week 16 | -6.08 (0.818) | -5.67 (0.852) | -6.17 (0.835) | -6.99 (0.836)

3. Secondary Outcome: Least Squares Mean Change From Baseline in ESSPRI Score at Week 24
Description: The EULAR Sjörgen's Syndrome Patient Reported Index (ESSPRI) is an established disease outcome measure for Sjögren's syndrome that is calculated by averaging the scales for pain, fatigue and dryness. The total score is the mean score of the 3 scales and ranges between 0 and 10 with higher values indicating more severity of symptoms. A negative change from baseline is a favorable outcome.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale | -1.71 (0.288) | -1.39 (0.304) | -1.70 (0.301) | -1.77 (0.295)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo; Test type: Superiority; p = 0.4457, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.32, 95% CI 2-sided [-0.50 to 1.13]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo; Test type: Superiority; p = 0.301, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Square Mean Difference = 0.01, 95% CI 2-sided [-0.79 to 0.82]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo; Test type: Superiority; p = 0.8858, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Square Mean Difference = -0.06, 95% CI 2-sided [-0.86 to 0.74]

4. Secondary Outcome: Least Squares Mean Change From Baseline in ESSPRI Score at Weeks 4, 8, 12 and 16
Description: as for outcome 3
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Week 4: number analyzed (Participants) | 48 | 46 | 46 | 46
  Week 4 | -0.54 (0.236) | -0.67 (0.247) | -0.80 (0.241) | -0.88 (0.242)
  Week 8: number analyzed (Participants) | 48 | 45 | 43 | 46
  Week 8 | -0.94 (0.242) | -0.84 (0.255) | -1.06 (0.251) | -1.8 (0.248)
  Week 12: number analyzed (Participants) | 48 | 44 | 45 | 47
  Week 12 | -1.42 (0.265) | -1.36 (0.279) | -1.44 (0.273) | -1.23 (0.270)
  Week 16: number analyzed (Participants) | 48 | 46 | 45 | 45
  Week 16 | -1.77 (0.263) | -1.27 (0.275) | -1.55 (0.271) | -1.55 (0.270)

5. Secondary Outcome: Least Squares Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) Score Over 24 Weeks
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F v4) is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during their usual daily activities over the previous week. The level of fatigue is measured on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The global score ranges between 0 and 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale | 9.05 (1.404) | 7.12 (1.502) | 6.48 (1.518) | 9.36 (1.436)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo; Test type: Superiority; p = 0.3424, Mixed Models Analysis; Confidence intervals and p-values are derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -1.93, 95% CI 2-sided [-5.93 to 2.07]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo; Test type: Superiority; p = 0.2092, Mixed Models Analysis; Confidence intervals and p-values are derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -2.56, 95% CI 2-sided [-6.58 to 1.45]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo; Test type: Superiority; p = 0.8740, Mixed Models Analysis; Confidence intervals and p-values are derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.31, 95% CI 2-sided [-3.58 to 4.20]

6. Secondary Outcome: Least Squares Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) Score at Weeks 4, 8, 12 and 16
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 48 | 42 | 39 | 46
Scores on a scale
  Week 4 | 3.78 (1.175) | 6.32 (1.239) | 3.12 (1.229) | 3.39 (1.203)
  Week 8 | 5.49 (1.222) | 6.36 (1.297) | 3.93 (1.303) | 5.98 (1.250)
  Week 12 | 6.25 (1.349) | 8.17 (1.429) | 5.73 (1.427) | 6.05 (1.374)
  Week 16 | 8.56 (1.284) | 7.09 (1.357) | 6.86 (1.359) | 8.30 (1.318)

7. Secondary Outcome: Least Squares Mean Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component (PCS) and Mental Component (MCS) Over 24 Weeks
Description: The SF36 includes 8 scale scores (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) and two summary scores, the physical and mental component scores. The first four and last four scales comprise physical and mental component scores, respectively. The range of scores of the physical component (PCS) and mental component (MCS) is 0 (lowest or worst possible level of functioning) to 100 (highest or best possible level of functioning).
Time Frame: Baseline, Week 24
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Mental Component Score: number analyzed (Participants) | 48 | 42 | 39 | 46
  Mental Component Score | 4.63 (1.259) | 3.61 (1.350) | 5.31 (1.367) | 5.63 (1.286)
  Physical Component Score: number analyzed (Participants) | 48 | 42 | 39 | 46
  Physical Component Score | 3.66 (0.952) | 4.79 (1.019) | 2.66 (1.026) | 5.50 (0.972)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo / Mental Component Score; Test type: Superiority; p = 0.5768, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -1.02, 95% CI 2-sided [-4.61 to 2.57]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo / Mental Component Score; Test type: Superiority; p = 0.7113, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.68, 95% CI 2-sided [-2.93 to 4.28]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo / Mental Component Score; Test type: Superiority; p = 0.5722, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 1.00, 95% CI 2-sided [-2.49 to 4.48]
Statistical Analysis 4: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo / Physical Component Score; Test type: Superiority; p = 0.4138, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 1.84, 95% CI 2-sided [-1.59 to 3.83]
Statistical Analysis 5: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo / Physical Component Score; Test type: Superiority; p = 0.4663, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -1.00, 95% CI 2-sided [-3.72 to 1.71]
Statistical Analysis 6: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo / Physical Component Score; Test type: Superiority; p = 0.1694, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 1.84, 95% CI 2-sided [-0.79 to 4.47]

8. Secondary Outcome: Least Squares Mean Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component (PCS) and Mental Component (MCS) at Weeks 4, 8, 12 and 16
Description: as for outcome 7
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: Full Analysis Set (FAS): Only participants with a value at both Baseline and post-baseline visit included.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Week 4 - Mental Component Score: number analyzed (Participants) | 48 | 45 | 44 | 46
  Week 4 - Mental Component Score | 0.49 (1.091) | 1.89 (1.151) | 2.46 (1.149) | 2.18 (1.116)
  Week 8 - Mental Component Score: number analyzed (Participants) | 48 | 44 | 41 | 46
  Week 8 - Mental Component Score | 2.65 (2.267) | 3.80 (1.341) | 4.65 (1.363) | 3.35 (1.294)
  Week 12 - Mental Component Score: number analyzed (Participants) | 48 | 44 | 43 | 47
  Week 12 - Mental Component Score | 2.89 (1.188) | 5.42 (1.264) | 3.94 (1.265) | 4.59 (1.207)
  Week 16 - Mental Component Score: number analyzed (Participants) | 48 | 45 | 43 | 45
  Week 16 - Mental Component Score | 4.60 (1.214) | 3.00 (1.281) | 5.57 (1.291) | 5.46 (1.247)
  Week 4 - Physical Component Score: number analyzed (Participants) | 48 | 45 | 44 | 46
  Week 4 - Physical Component Score | 3.35 (0.844) | 3.94 (0.889) | 1.14 (0.878) | 1.98 (0.863)
  Week 8 - Physical Component Score: number analyzed (Participants) | 48 | 44 | 43 | 47
  Week 8 - Physical Component Score | 3.83 (0.894) | 4.56 (0.949) | 3.48 (0.941) | 3.47 (0.909)
  Week 12 - Physical Component Score: number analyzed (Participants) | 48 | 44 | 43 | 47
  Week 12 - Physical Component Score | 3.83 (0.894) | 4.56 (0.949) | 3.48 (0.941) | 3.47 (0.909)
  Week 16 - Physical Component Score: number analyzed (Participants) | 48 | 45 | 43 | 45
  Week 16 - Physical Component Score | 4.72 (0.968) | 4.67 (1.020) | 3.32 (1.021) | 4.57 (0.993)

9. Secondary Outcome: Least Squares Mean Change From Baseline in Physician's Global Assessment (PhGA) of Patient's Overall Disease Activity Using Patient Visual Analog Scale (VAS) Over 24 Weeks
Description: Physician global assessment of overall disease activity (PhGA) was performed using a 100 mm visual analogue scale (VAS) ranging from no disease activity (score 0) to maximal disease activity (score 100), after the question "Considering all the ways the disease affects your patient, draw a line on the scale for how well his or her condition is today". A negative change from baseline is a favourable outcome.
Time Frame: Baseline, 24 weeks
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale | -23.64 (2.601) | -27.81 (2.751) | -28.13 (2.700) | -31.99 (2.630)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo; Test type: Superiority; p = 0.2671, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -4.17, 95% CI 2-sided [-11.56 to 3.22]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo; Test type: Superiority; p = 0.2248, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -4.49, 95% CI 2-sided [-11.78 to 2.79]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo; Test type: Superiority; p = 0.0224, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -8.36, 95% CI 2-sided [-15.51 to -1.20]

10. Secondary Outcome: Least Squares Mean Change From Baseline in Physician's Global Assessment (PhGA) of Patient's Overall Disease Activity Using Patient Visual Analog Scale (VAS) at Weeks 4, 8, 12 and 16
Description: as for outcome 9
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Week 4: number analyzed (Participants) | 47 | 43 | 45 | 45
  Week 4 | -12.49 (2.327) | -10.50 (2.445) | -12.38 (2.361) | -18.67 (2.367)
  Week 8: number analyzed (Participants) | 48 | 45 | 40 | 45
  Week 8 | -18.54 (2.239) | -16.53 (2.338) | -22.12 (2.374) | -24.85 (2.289)
  Week 12 | -21.01 (2.299) | -20.72 (2.413) | -25.35 (2.341) | -27.25 (2.305)
  Week 16 | -19.44 (2.572) | -24.49 (2.687) | -24.77 (2.676) | -25.77 (2.633)

11. Secondary Outcome: Patient's Global Assessment (PaGA) Score at Weeks 4, 8, 12, 16 and 24
Description: The PaGA of disease activity was performed using a 100 mm Visual Analog Scale (VAS) ranging from 0 (no disease activity) to 100 (maximal disease activity), in response to the question "Considering all the ways Sjögren's syndrome affects you, please draw a line on the scale to indicate how well you are doing today". A negative change from baseline is a favourable outcome.
Time Frame: Weeks 4, 8, 12, 16 and 24
Population: Full Analysis Set (FAS). Only participants with a value at both Baseline and post-baseline visit included.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
Scores on a scale
  Week 4: number analyzed (Participants) | 48 | 45 | 44 | 46
  Week 4 | -9.42 (2.850) | -10.02 (2.992) | -5.96 (2.969) | -8.96 (2.906)
  Week 8: number analyzed (Participants) | 48 | 44 | 40 | 46
  Week 8 | -9.74 (3.035) | -11.48 (3.214) | -8.70 (3.271) | -15.27 (3.091)
  Week 12: number analyzed (Participants) | 48 | 44 | 43 | 47
  Week 12 | -11.45 (3.064) | -17.51 (3.244) | -11.73 (3.234) | -13.57 (3.105)
  Week 16 | -16.26 (3.194) | -17.56 (3.361) | -14.86 (3.375) | -15.78 (3.271)
  Week 24 | -15.11 (3.405) | -12.83 (3.648) | -11.85 (3.704) | -19.87 (3.470)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo; Test type: Superiority; p = 0.6457, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 2.27, 95% CI 2-sided [-7.46 to 12.00]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo; Test type: Superiority; p = 0.5132, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 3.26, 95% CI 2-sided [-6.55 to 13.06]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo; Test type: Superiority; p = 95, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -4.77, 95% CI 2-sided [-14.21 to 4.68]

12. Secondary Outcome: Least Squares Mean Change From Baseline in Salivary Flow Rate at Week 24
Description: Change from baseline in salivary flow rate (unstimulated and stimulated) at 24 weeks as compared to placebo.
  Unstimulated saliva is a mix of serous and mucous secretions coming primarily from the submandibular and minor salivary glands. The parotid gland produces the largest volume of stimulated saliva. Stimulated saliva accounts for 80-90% of daily salivary production.
Time Frame: Baseline, 24 weeks
Population: Full analysis set (FAS): The overall number of participants analyzed represents the FAS. The number analyzed per row represents participants with data available at each assessment.
Measure: Least Squares Mean (Standard Error); unit: mL/min
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24)
Number analyzed (Participants) | 49 | 47 | 47 | 47
mL/min
  Stimulated: number analyzed (Participants) | 47 | 40 | 41 | 45
  Stimulated | 0.05 (0.067) | 0.16 (0.074) | 0.18 (0.071) | 0.25 (0.98)
  Unstimulated: number analyzed (Participants) | 46 | 38 | 41 | 45
  Unstimulated | 0.00 (0.030) | 0.01 (0.034) | -0.00 (0.032) | -0.01 (0.031)
Statistical Analysis 1: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo (Stimulated salivary flow rate); Test type: Superiority; p = 0.2710, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.08 to 0.30]
Statistical Analysis 2: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo (Stimulated salivary flow rate); Test type: Superiority; p = 0.1618, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.13, 95% CI 2-sided [-0.05 to 0.32]
Statistical Analysis 3: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo (Stimulated salivary flow rate); Test type: Superiority; p = 0.0374, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.20, 95% CI 2-sided [0.01 to 0.38]
Statistical Analysis 4: Comparison: Placebo (Up to Week 24) vs VAY736 - 5 mg (Up to Week 24); Week 24: VAY736 5 mg vs. Placebo (Unstimulated salivary flow rate); Test type: Superiority; p = 0.9559, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = 0.00, 95% CI 2-sided [-0.09 to 0.09]
Statistical Analysis 5: Comparison: Placebo (Up to Week 24) vs VAY736 - 50 mg (Up to Week 24); Week 24: VAY736 50 mg vs. Placebo (Unstimulated salivary flow rate); Test type: Superiority; p = 0.9290, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -0.00, 95% CI 2-sided [-0.09 to 0.08]
Statistical Analysis 6: Comparison: Placebo (Up to Week 24) vs VAY736 - 300 mg (Up to Week 24); Week 24: VAY736 300 mg vs. Placebo (Unstimulated salivary flow rate); Test type: Superiority; p = 0.7276, Mixed Models Analysis; Confidence intervals and p-values derived from a mixed model for repeated measures (MMRM); Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.10 to 0.07]

13. Secondary Outcome: Percent Change From Baseline in Whole Blood CD19+ B-cell Counts.
Description: B-cell counts were measured before, during and after treatment with VAY736. After stopping VAY736 treatment they were used to monitor patients for time to recovery of adequate CD19+ B cell counts prior to discharge from the study. Change from baseline in B-cell counts before, during and after treatment with VAY736 as well as the time to recover to baseline like values (defined as at least 80% of baseline counts or >= 50 cells/μL) were analyzed by descriptive statistics.
  Baseline was defined as the last assessment performed on or prior to the date of administration of the first dose of study treatment.
Time Frame: Baseline, Week 24, Week 28
Population: Full analysis set (FAS): patients were analyzed according to the first treatment received (at Period 2, 24 weeks). VAY736 300 mg - Placebo included patients who discontinued in Period 2 and entered Period 4 directly and patients who completed Period 2 and were re-randomized to placebo. Only patients with baseline measurement and at least one measurement post-baseline were included.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo - VAY150 mg: Placebo control at 24 weeks VAY150g at 28 weeks
Arm/Group | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | Placebo - VAY150 mg | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Number analyzed (Participants) | 47 | 47 | 49 | 26 | 21
Percent change
  Week 24: number analyzed (Participants) | 35 | 34 | 36 | 17 | 18
  Week 24 | -88.00 (5.784) | -99.07 (5.812) | 3.29 (5.674) | -103.0 (8.198) | -94.20 (8.098)
  Week 28: number analyzed (Participants) | 0 | 0 | 35 | 13 | 17
  Week 28 |  |  | -97.06 (5.732) | -105.3 (9.145) | -91.80 (8.272)

14. Secondary Outcome: Kaplan-Meier Analysis for Time to Recovery to Baseline Like Values for B-cell Counts
Description: as for outcome 13
Time Frame: Up to two years from last dose patient received.
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Placebo - VAY150 mg: Placebo control at week 24 VAY150 mg at week 28
Arm/Group | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | Placebo - VAY150 mg | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Number analyzed (Participants) | 47 | 47 | 49 | 26 | 21
months | 3.8 [2.7 to 5.2] | 4.8 [4.7 to 6.6] | 6.8 [5.0 to 9.2] | 8.4 [6.8 to 9.1] | 6.5 [4.9 to 7.5]

15. Secondary Outcome: Peak Serum Concentration of VAY736
Description: Pharmacokinetic Concentrations
  This outcome only applies to patients who received at least one dose of VAY739 (so not applicable to placebo)
Time Frame: baseline to week 24, then week 28
Population: Safety set (SAF): included all patients who received at least one dose of study medication. Patients were analyzed according to treatment received and the actual stratum at baseline. The safety set was used in the analysis of all safety variables.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | VAY736 300 mg - Placebo | VAY736 300 mg - VAY736 300 mg
Number analyzed (Participants) | 47 | 47 | 4 | 21 | 22
ug/mL | 0.0747 (0.203) | 0.475 (0.380) | 1.46 (0.596) | 2.15 (1.47) | 1.94 (1.53)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of follow-up period, up to approximately 3 years (max duration of follow-up was 2 years).
Description: An adverse event is any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Groups:
- Any VAY736 (Up to Week 24); ALL (Up to Week 24): Period 2 (Double blind Placebo s.c. administration every 4 weeks (q4w) for a 24-week period)
- VAY736 - 5 mg 24 Weeks (Periods 2 and 4): All events reported from start of VAY736 - 5 mg dose in Period 2 (blinded treatment period of 24 weeks) and in the post treatment safety follow-up (Period 4)
- VAY736 - 50 mg 24 Weeks (Periods 2 and 4): All events reported from start of VAY736 - 50 mg dose in Period 2 (blinded treatment period of 24 weeks) and in the post treatment safety follow-up (Period 4)
- VAY736 - 150 mg 28 Weeks (Periods 3 and 4): All events reported from start of VAY736 - 150 mg dose in Period 3 (extended blinded treatment period of 28 weeks) up to the end of post treatment safety follow-up (Period 4)
- VAY736 - 300 mg 24 Weeks (Entire Study); VAY736 - 300 mg 52 Weeks (Entire Study); Any VAY736 - 300 mg (Periods 2, 3 and 4); Any VAY736 (Periods 2, 3 and 4): All events reported from the beginning of the study up until the end of post treatment safety follow-up (Period 4)
Arm/Group | Placebo (Up to Week 24) | VAY736 - 5 mg (Up to Week 24) | VAY736 - 50 mg (Up to Week 24) | VAY736 - 300 mg (Up to Week 24) | Any VAY736 (Up to Week 24) | ALL (Up to Week 24) | VAY736 - 5 mg 24 Weeks (Periods 2 and 4) | VAY736 - 50 mg 24 Weeks (Periods 2 and 4) | VAY736 - 150 mg 28 Weeks (Periods 3 and 4) | VAY736 - 300 mg 24 Weeks (Entire Study) | VAY736 - 300 mg 52 Weeks (Entire Study) | Any VAY736 - 300 mg (Periods 2, 3 and 4) | Any VAY736 (Periods 2, 3 and 4)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47 | 0/47 | 0/47 | 0/141 | 0/190 | 0/47 | 0/47 | 0/47 | 0/26 | 0/21 | 0/47 | 0/188
Serious Adverse Events (participants affected / at risk) | 3/49 | 0/47 | 1/47 | 2/47 | 3/141 | 6/190 | 3/47 | 7/47 | 9/47 | 5/26 | 5/21 | 10/47 | 29/188
Other Adverse Events (participants affected / at risk) | 33/49 | 40/47 | 34/47 | 41/47 | 115/141 | 148/190 | 41/47 | 37/47 | 41/47 | 24/26 | 20/21 | 44/47 | 163/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to Week 24) (N=49) | VAY736 - 5 mg (Up to Week 24) (N=47) | VAY736 - 50 mg (Up to Week 24) (N=47) | VAY736 - 300 mg (Up to Week 24) (N=47) | Any VAY736 (Up to Week 24) (N=141) | ALL (Up to Week 24) (N=190) | VAY736 - 5 mg 24 Weeks (Periods 2 and 4) (N=47) | VAY736 - 50 mg 24 Weeks (Periods 2 and 4) (N=47) | VAY736 - 150 mg 28 Weeks (Periods 3 and 4) (N=47) | VAY736 - 300 mg 24 Weeks (Entire Study) (N=26) | VAY736 - 300 mg 52 Weeks (Entire Study) (N=21) | Any VAY736 - 300 mg (Periods 2, 3 and 4) (N=47) | Any VAY736 (Periods 2, 3 and 4) (N=188)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Cell-mediated immune deficiency (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to Week 24) (N=49) | VAY736 - 5 mg (Up to Week 24) (N=47) | VAY736 - 50 mg (Up to Week 24) (N=47) | VAY736 - 300 mg (Up to Week 24) (N=47) | Any VAY736 (Up to Week 24) (N=141) | ALL (Up to Week 24) (N=190) | VAY736 - 5 mg 24 Weeks (Periods 2 and 4) (N=47) | VAY736 - 50 mg 24 Weeks (Periods 2 and 4) (N=47) | VAY736 - 150 mg 28 Weeks (Periods 3 and 4) (N=47) | VAY736 - 300 mg 24 Weeks (Entire Study) (N=26) | VAY736 - 300 mg 52 Weeks (Entire Study) (N=21) | Any VAY736 - 300 mg (Periods 2, 3 and 4) (N=47) | Any VAY736 (Periods 2, 3 and 4) (N=188)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 6 | 11 | 13 | 3 | 2 | 4 | 2 | 4 | 6 | 15
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2 | 4 | 2 | 8 | 11 | 4 | 4 | 3 | 1 | 1 | 2 | 13
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 4 | 8 | 9 | 5 | 1 | 2 | 2 | 2 | 4 | 12
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 2 | 3 | 1 | 1 | 1 | 0 | 2 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 3 | 8 | 12 | 3 | 3 | 2 | 3 | 4 | 7 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 5 | 6 | 1 | 4 | 0 | 0 | 1 | 1 | 6
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 2 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 4 | 4 | 1 | 1 | 1 | 2 | 0 | 2 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Influenza like illness (General disorders) | 1 | 0 | 3 | 1 | 4 | 5 | 0 | 4 | 1 | 2 | 2 | 4 | 9
Injection site reaction (General disorders) | 2 | 4 | 9 | 26 | 39 | 41 | 4 | 9 | 17 | 13 | 14 | 27 | 57
Oedema peripheral (General disorders) | 2 | 0 | 2 | 2 | 4 | 6 | 0 | 2 | 0 | 2 | 1 | 3 | 5
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 3 | 3 | 0 | 3 | 7
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 0 | 2 | 0 | 1 | 1 | 6
Bronchitis (Infections and infestations) | 2 | 3 | 2 | 2 | 7 | 9 | 3 | 3 | 4 | 2 | 2 | 4 | 14
Conjunctivitis (Infections and infestations) | 3 | 3 | 2 | 2 | 7 | 10 | 3 | 5 | 2 | 2 | 0 | 2 | 12
Cystitis (Infections and infestations) | 0 | 0 | 1 | 2 | 3 | 3 | 0 | 1 | 2 | 2 | 1 | 3 | 6
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 1 | 3 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 7
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 4 | 5
Nasopharyngitis (Infections and infestations) | 5 | 4 | 2 | 7 | 13 | 18 | 7 | 4 | 11 | 5 | 4 | 9 | 31
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 4
Oral herpes (Infections and infestations) | 1 | 3 | 1 | 0 | 4 | 5 | 4 | 2 | 2 | 1 | 3 | 4 | 12
Parotitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 1 | 0 | 1 | 6
Sinusitis (Infections and infestations) | 4 | 4 | 2 | 0 | 6 | 10 | 5 | 3 | 7 | 2 | 1 | 3 | 18
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 3 | 4 | 4 | 1 | 0 | 0 | 1 | 2 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 5 | 2 | 11 | 15 | 7 | 9 | 7 | 8 | 2 | 10 | 33
Urinary tract infection (Infections and infestations) | 4 | 6 | 2 | 0 | 8 | 12 | 9 | 5 | 7 | 2 | 3 | 5 | 26
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 3 | 3 | 1 | 1 | 0 | 2 | 0 | 2 | 4
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 2 | 2 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 3 | 5
Injection related reaction (Injury, poisoning and procedural complications) | 2 | 6 | 5 | 4 | 15 | 17 | 6 | 5 | 7 | 2 | 2 | 4 | 22
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 3
Blood creatinine increased (Investigations) | 2 | 2 | 1 | 0 | 3 | 5 | 3 | 1 | 1 | 1 | 0 | 1 | 6
Lymphocyte count decreased (Investigations) | 0 | 4 | 0 | 0 | 4 | 4 | 4 | 0 | 1 | 0 | 2 | 2 | 7
Neutrophil count decreased (Investigations) | 0 | 3 | 0 | 0 | 3 | 3 | 3 | 0 | 1 | 1 | 1 | 2 | 6
White blood cell count decreased (Investigations) | 1 | 3 | 1 | 1 | 5 | 6 | 3 | 1 | 0 | 1 | 1 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 1 | 5 | 10 | 3 | 1 | 6 | 2 | 3 | 5 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 2 | 7 | 10 | 3 | 4 | 6 | 4 | 2 | 6 | 19
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 3 | 4 | 2 | 0 | 0 | 2 | 1 | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 2 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 3 | 4 | 2 | 0 | 4 | 1 | 2 | 3 | 9
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 4 | 4 | 3 | 4 | 2 | 2 | 0 | 2 | 11
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 2 | 2 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 3 | 4 | 4 | 2 | 1 | 0 | 2 | 2 | 4 | 7
Headache (Nervous system disorders) | 7 | 4 | 4 | 4 | 12 | 19 | 5 | 5 | 4 | 4 | 2 | 6 | 20
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 3 | 0 | 3 | 3 | 6
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 4 | 5 | 3 | 0 | 2 | 2 | 0 | 2 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 4 | 5 | 2 | 1 | 2 | 2 | 1 | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 1 | 7 | 10 | 6 | 3 | 2 | 2 | 2 | 4 | 15
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 3 | 3 | 4 | 2 | 2 | 0 | 0 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT02962895/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02962895/SAP_001.pdf